CLINICAL TRIAL: NCT00136955
Title: An Open Labeled, Single-Arm, Multicentre Phase II Study To Evaluate The Efficacy And Safety Of Weekly Irinotecan Plus Cisplatin As First-Line Chemotherapy For Advanced Or Recurrent Squamous Cell Carcinoma Of The Uterine Cervix
Brief Title: Irinotecan Study For Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XRP4174/2502; A5961083
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Results first posted 2009-06-25 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-05

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Weekly Irinotecan(60mg/sqm, D1, 8, 15) in combination with Cisplatin (60mg/sqm, D1), Squamous Cell Carcinoma Of The Uterine Cervix
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- irinitecan/cisplatin (Experimental): experimental arm consists of patients who receive irinotecan/cisplatin
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Irinotecan — An Open Labeled, Single-Arm, Multicentre Phase II Study To Evaluate The Efficacy And Safety Of Weekly Irinotecan (60mg/sqm, D1, 8, 15) Plus Cisplatin (60mg/sqm, D1) As First-Line Chemotherapy For Advanced Or Recurrent Squamous Cell Carcinoma Of The Uterine Cervix

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of Irinotecan plus cisplatin as first-line chemotherapy for advanced or recurrent cervical cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented, advanced or recurrent squamous cell carcinoma of uterine cervix. Patients may have received concurrent (with radiotherapy) or (neo)adjuvant (before or after local treatment) chemotherapy for primary tumor providing that at least 6 months have passed from the completion of previous therapy and the diagnosis of recurrent disease was documented
* Having measurable lesion(s), without previous radiation therapy.

Exclusion Criteria:

* Patients had ever received primary chemotherapy for cervical cancer other than mentioned previously (in the inclusion criteria).
* Patients ever received cisplatin with total dose > 300 mg/m2 and received radiotherapy or local treatment delivered to the target lesion.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2004-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Taiwan (5):
  - Pfizer Investigational Site, Kwei-Shan County, TaoYuan,, Taiwan
  - Pfizer Investigational Site, Taichung, Taiwan
  - Pfizer Investigational Site, Taipei, Taiwan
  - Pfizer Investigational Site, Kaoshiung
  - Pfizer Investigational Site, Taipei

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=XRP4174/2502&StudyName=Irinotecan%20Study%20For%20Cervical%20Cancer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 41 subjects had a primary diagnosis of squamous cell carcinoma of the cervix with a mean duration of 2.8 years (range: 0-12.9 years) since first diagnosis. No subject had a history of other cancer.
Groups:
- Irinotecan/Cisplatin: Intravenous irinotecan (60 milligrams [mg]/metered square [m2]) on days 1, 8, and 15 plus cisplatin (60mg/m2) on day 1. Treatment cycle was repeated every 4 weeks.
Period: Overall Study
Arm/Group | Irinotecan/Cisplatin
Started | 41
Completed | 18
Not Completed | 23
Not completed — Adverse Event | 8
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2
Not completed — Incl. prog. disease, protocol violation | 12

BASELINE CHARACTERISTICS:
Arm/Group | Irinotecan/Cisplatin
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Response to Treatment Based on Response Evaluation Criteria in Solid Tumors (RECIST) Criteria (Evaluable Population)
Description: Tumor response according to RECIST.
Time Frame: At baseline and every 8 weeks through end of treatment (21-28 days after last administration of study treatment)
Population: Evaluable population: 1) Patient received at least two complete cycles of treatment (8 weeks on study). If progression occurred before end of second cycle, patient considered evaluable (early progression); 2) all baseline lesions assessed at least once after second cycle with same method of measurement as baseline; 3) no major protocol violation.
Measure: Number; unit: participant
Arm/Group | Irinotecan/Cisplatin
Number analyzed (Participants) | 32
participant
  complete response (CR) | 8
  partial response (PR) | 7
  stable disease (SD) | 11
  progressive disease (PD) | 6
  not evaluable | 0
  missing | 0
  Response Rate (PR + CR) - naive | 15
  Response Rate (PR + CR) - corrected | 15

2. Secondary Outcome: Overall Survival (OS) and Time to Tumor Progression (TTP) (Evaluable Population)
Description: TTP is date of first infusion to first date of documented progression or date of death due to progressive disease or date of further anti-tumor therapy, whichever occurs first. OS is time from date of first infusion to date of death due to any cause or last date patient is known to be alive at date of data cutoff for final analysis.
Time Frame: Tumor response measurements were made at baseline, according to RECIST criteria. After end of treatment, subject was followed-up every 12 weeks plus or minus 2 weeks.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Irinotecan/Cisplatin
Number analyzed (Participants) | 32
days
  Overall Survival | 652 [398 to 840]
  Time to tumor progression | 277 [157 to 682]

3. Primary Outcome: Response to Treatment Based on RECIST Criteria (Intent-to-Treat [ITT] Population)
Description: Tumor response according to RECIST.
Time Frame: At baseline and every 8 weeks through end of treatment (21-28 days after last administration of study treatment)
Population: Intent-to-treat (ITT) population: All included subjects who received at least one drop of study medication will be included in the ITT population.
Measure: Number; unit: participant
Arm/Group | Irinotecan/Cisplatin
Number analyzed (Participants) | 41
participant
  complete response | 8
  partial response | 8
  stable disease | 13
  progressive disease | 8
  not evaluable | 4
  missing | 0
  Response Rate (PR + CR) - naive | 16

4. Secondary Outcome: Overall Survival (OS) and Time to Tumor Progression (ITT Population)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Irinotecan/Cisplatin
Number analyzed (Participants) | 41
days
  Overall Survival | 448 [348 to 680]
  Time to Tumor Progression | 263 [157 to 652]

ADVERSE EVENTS:
Arm/Group | Irinotecan/Cisplatin
Serious Adverse Events (participants affected / at risk) | 25
Other Adverse Events (participants affected / at risk) | 40
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Irinotecan/Cisplatin
Febrile neutropenia (Blood and lymphatic system disorders) | 3/41
Leukopenia (Blood and lymphatic system disorders) | 14/41
Diarrhoea (Gastrointestinal disorders) | 6/41
Gastrointestinal disorder (Gastrointestinal disorders) | 1/41
Ileus (Gastrointestinal disorders) | 1/41
Nausea (Gastrointestinal disorders) | 5/41
Proctitis (Gastrointestinal disorders) | 1/41
Vomiting (Gastrointestinal disorders) | 5/41
Asthenia (General disorders) | 4/41
Pyrexia (General disorders) | 8/41
Infection (Infections and infestations) | 10/41
Haemoglobin (Investigations) | 9/41
Neutrophil count decreased (Investigations) | 13/41
Platelet count (Investigations) | 4/41
Weight decreased (Investigations) | 1/41
Anorexia (Metabolism and nutrition disorders) | 2/41
Hypercalcaemia (Metabolism and nutrition disorders) | 1/41
Hypokalaemia (Metabolism and nutrition disorders) | 1/41
Depressed level of consciousness (Nervous system disorders) | 1/41
Syncope (Nervous system disorders) | 1/41
Bladder pain (Renal and urinary disorders) | 1/41
Urinary retention (Renal and urinary disorders) | 1/41
Urogenital disorder (Renal and urinary disorders) | 1/41
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/41
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1/41
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1/41
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1/41
Skin disorder (Skin and subcutaneous tissue disorders) | 1/41
Hypotension (Vascular disorders) | 2/41
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Irinotecan/Cisplatin
Blood disorder (Blood and lymphatic system disorders) | 9/41
Leukopenia (Blood and lymphatic system disorders) | 24/41
Abdominal pain (Gastrointestinal disorders) | 6/41
Constipation (Gastrointestinal disorders) | 7/41
Diarrhoea (Gastrointestinal disorders) | 26/41
Flatulence (Gastrointestinal disorders) | 3/41
Gastrointestinal disorder (Gastrointestinal disorders) | 3/41
Nausea (Gastrointestinal disorders) | 20/41
Vomiting (Gastrointestinal disorders) | 27/41
Asthenia (General disorders) | 10/41
Oedema (General disorders) | 3/41
Pain (General disorders) | 10/41
Pyrexia (General disorders) | 3/41
Infection (Infections and infestations) | 11/41
Alanine aminotransferase increased (Investigations) | 3/41
Aspartate aminotransferase increased (Investigations) | 4/41
Haemoglobin (Investigations) | 32/41
Neutrophil count decreased (Investigations) | 16/41
Platelet count (Investigations) | 15/41
Weight decreased (Investigations) | 5/41
Anorexia (Metabolism and nutrition disorders) | 10/41
Dizziness (Nervous system disorders) | 4/41
Headache (Nervous system disorders) | 3/41
Insomnia (Psychiatric disorders) | 10/41
Micturition disorder (Renal and urinary disorders) | 3/41
Renal failure (Renal and urinary disorders) | 4/41
Urinary retention (Renal and urinary disorders) | 3/41
Vaginal haemorrhage (Reproductive system and breast disorders) | 4/41
Cough (Respiratory, thoracic and mediastinal disorders) | 10/41
Alopecia (Skin and subcutaneous tissue disorders) | 10/41
Exfoliative rash (Skin and subcutaneous tissue disorders) | 4/41
Pruritus (Skin and subcutaneous tissue disorders) | 3/41
Skin disorder (Skin and subcutaneous tissue disorders) | 3/41
Packed red blood cell transfusion (Surgical and medical procedures) | 5/41
Hypertension (Vascular disorders) | 4/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.